CLINICAL TRIAL: NCT05475548
Title: Effect of Skeletally Anchored Reversed PowerScope Appliance in Orthodontic Treatment of Patients With Class III Malocclusion: A Prospective Clinical Study
Brief Title: Effect of Skeletally Anchored Reversed PowerScope Appliance in Orthodontic Treatment of Patients With Class III Malocclusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ibrahim Sallam, principal investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 786/2231
Record Dates: First submitted 2022-07-17; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Effect of PowerScope Appliance in Treatment of Patients With Class 3 Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): using reversed skeletally anchored PowerScope as a fixed functional appliance. (Active Comparator): eight patients with mild to moderate Class IΙΙ malocclusion who will be treated by pre-adjusted straight wire appliance followed by reversed skeletally anchored PowerScope as a fixed functional appliance.
  Interventions: Device: powerscope
- Group (B): using dentally anchored reversed PowerScope as a fixed functional appliance (Active Comparator): eight patients with mild to moderate Class IΙΙ malocclusion who will be treated by pre-adjusted straight wire appliance followed by dentally anchored reversed PowerScope as a fixed functional appliance
  Interventions: Device: powerscope

INTERVENTIONS:
Device: powerscope — The PowerScope is the latest innovation in the treatment of Class II malocclusion which is a direct derivative of the Herbst Type II appliance. Dr. Andy Hayes worked in conjunction with American Orthodontics to develop PowerScope in 2016. This appliance supports intermaxillary wire-to-wire installation via a nut and hexagonal screw. A ball and socket joint is used to maximize lateral movement while improving patient comfort. The appliance is made up of a telescopic mechanism made up of an inner shaft/push rod, middle and outer tubing, and a spacer between the middle and outer tubing. A nickel-titanium (NiTi) spring provides a constant 260 g force. According to the present knowledge no studies regarding treatment outcomes of comprehensive fixed appliance treatment combined with the PowerScope in Class ΙII patients have been reported

SUMMARY:
the PowerScope appliance is found to be efficient for the treatment of class II malocclusion. Accordingly, it appears valuable to investigate the efficiency of skeletally anchored powerScope in the treatment of class III malocclusion

DETAILED DESCRIPTION:
The PowerScope is the latest innovation in the treatment of Class II malocclusion which is a direct derivative of the Herbst Type II appliance. Dr. Andy Hayes worked in conjunction with American Orthodontics to develop PowerScope in 2016. This appliance supports intermaxillary wire-to-wire installation via a nut and hexagonal screw. A ball and socket joint is used to maximize lateral movement while improving patient comfort. The appliance is made up of a telescopic mechanism made up of an inner shaft/push rod, middle and outer tubing, and a spacer between the middle and outer tubing. A nickel-titanium (NiTi) spring provides a constant 260 g force. According to the present knowledge no studies regarding treatment outcomes of comprehensive fixed appliance treatment combined with the PowerScope in Class ΙII patients have been reported.

The introduction of temporary anchorage devices (TADs) has made it possible to achieve absolute anchorage control in daily clinical orthodontic practice when used in conjunction with fixed functional appliances. However, it appears that there is no evidence in the literature supporting the clinical effectiveness of miniscrew- anchored fixed functional appliances for the treatment of Class III malocclusion.

According to the current available literature, the PowerScope appliance is found to be efficient for the treatment of class II malocclusion. Accordingly, it appears valuable to investigate the efficiency of skeletally anchored powerScope in the treatment of class III malocclusion.

ELIGIBILITY:
Inclusion Criteria :

1. Mild to moderate Class III malocclusion adolescent patients with ANB (-3 - 0).
2. All permanent teeth are erupted (3rd molar not included).
3. An age of patients range from 14 to 18 years.
4. Good oral and general health.
5. No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement.
6. No previous orthodontic treatment.

Exclusion Criteria:

1. Orthodontic cases with severe crowding of upper and lower anterior segment that require extraction treatment approach.
2. Patients with a blocked-out tooth that will not allow for placement of the bracket at the initial bonding appointment.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of different dentoskeletal cephalometric parameters | 1.5 years
  amount of dentoskeletal change by cephalometric
Evaluation soft tissue parameters | 1.5 years
  amount of soft tissue change by cephalometric

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Sallam, student, Principal Investigator — Al-Azhar University
Locations (1):
- Ahmed Mohamed Ibrahim Sallam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of treatment for Class II malocclusion with the Herbst or twin-block appliances: a randomized, controlled trial. Am J Orthod Dentofacial Orthop. 2003 Aug;124(2):128-37. doi: 10.1016/s0889-5406(03)00345-7. PMID 12923506
- [Background] Eissa O, El-Shennawy M, Gaballah S, El-Meehy G, El Bialy T. Treatment outcomes of Class II malocclusion cases treated with miniscrew-anchored Forsus Fatigue Resistant Device: A randomized controlled trial. Angle Orthod. 2017 Nov;87(6):824-833. doi: 10.2319/032717-214.1. Epub 2017 Sep 8. PMID 28885034